CLINICAL TRIAL: NCT01470755
Title: Study on Dose-response to Bronchodilator Then Bronchodilator Dose-finding Using the Flow Interruption Technique in Children Aged 2.5 TO 6 Years
Brief Title: Study of Dose-response to Bronchodilator and Dose-finding in Child 2.5 to 6 Years - Study Golden
Acronym: DORESI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P100504; 2011-002261-38 (EudraCT Number)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2011-07

CONDITIONS: Asthma
Keywords: Pediatrics; Bronchial wheeze; bronchodilator; lung function; airway resistance
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- salbutamol - dose 1 (Other): Metered dose inhaler, 100µg+300µg per puff, administered one day
  Interventions: Drug: salbutamol
- Salbutamol - dose2 (Other): Metered dose inhaler, 100µg+500µg per puff, administered one day
  Interventions: Drug: Salbutamol - dose2
- Salbutamol - dose3 (Other): Metered dose inhaler, 200µg+600µg per puff, administered one day
  Interventions: Drug: Salbutamol -dose3
- salbutamol - dose4 (Other): Metered dose inhaler, 200µg+200µg per puff, administered one day
  Interventions: Drug: salbutamol -dose4

INTERVENTIONS:
Drug: salbutamol — Metered dose inhaler, 100µg+300µg per puff, administered one day
  Other Names: Salbutamol -100µg+300µg
  Arms: salbutamol - dose 1
Drug: Salbutamol - dose2 — Metered dose inhaler, 100µg+500µg per puff, administered one day
  Other Names: salbutamol -100µg+500µg
  Arms: Salbutamol - dose2
Drug: Salbutamol -dose3 — Metered dose inhaler, 200µg+600µg per puff, administered one day
  Other Names: salbutamol -200µg+600µg
  Arms: Salbutamol - dose3
Drug: salbutamol -dose4 — Metered dose inhaler, 200µg+200µg per puff, administered one day
  Other Names: salbutamol -200µg+200µg
  Arms: salbutamol - dose4

SUMMARY:
In older children and adults, bronchodilator (BD) dose-effect relationship is part of the characteristics of asthma disease. There are no data on BD dose-response relationship in wheezy preschool children whose disease pathophysiology is poorly understood, but may, in part, takes on the characteristics of asthma.

The investigators assume that 1) in young children interrupter resistance (Rint) could be used to measure a BD effect 2) the response to BD may vary depending on the dose used 3) the dose-response relationship could depend on the environment and gene polymorphism ADBR2.

This is a prospective phase II study on dose-response relationship and description of the dose-response curve design using a "sparse" and a modeling approach MCP-Mod.

The dose-response relationship will be modeled by sparse data. The investigators will test two doses per child in four designs that will be drawn. These doses will be assessed using Rint technique by a person blinded to the actual dose delivered to the child.

Measurements of 90 children will estimate E0, Imax and D50 (pharmacokinetic constants) with an accuracy of 3.5%, 8.9% and 25.7% respectively.

The bronchodilator used in the study is the Salbutamol as Ventolin ® (GSK) suspension for inhalation as an aerosol at a dose of 100μg per puff. Ventolin ® is used as part of the MA (No. 344 387-3)

DETAILED DESCRIPTION:
In older children and adults, bronchodilator (BD) dose-effect relationship is part of the characteristics of asthma disease. There are no data on BD dose-response relationship in wheezy preschool children whose disease pathophysiology is poorly understood, but may, in part, takes on the characteristics of asthma.

We assume that 1) in young children interrupter resistance (Rint) could be used to measure a BD effect 2) the response to BD may vary depending on the dose used 3) the dose-response relationship could depend on the environment and gene polymorphism ADBR2.

This is a prospective phase II study on dose-response relationship and description of the dose-response curve design using a "sparse" and a modeling approach MCP-Mod.

The dose-response relationship will be modeled by sparse data. We will test two doses per child in four designs that will be drawn. These doses will be assessed using Rint technique by a person blinded to the actual dose delivered to the child.

Measurements of 90 children will estimate E0, Imax and D50 (pharmacokinetic constants) with an accuracy of 3.5%, 8.9% and 25.7% respectively.

The bronchodilator used in the study is the Salbutamol as Ventolin ® (GSK) suspension for inhalation as an aerosol at a dose of 100μg per puff. Ventolin ® is used as part of the MA (No. 344 387-3) clinical implications The demonstration, first, of the possibility for Rint to detect a dose-response to BD will lead, secondly, to the determination of the minimum dose required for the detection of a reversibility in young children using Rint. It will end a long-standing debate about whether, when no Rint change is observed after BD administration in a young child, the child has actually no reversibility or the BD dose used was not sufficient to demonstrate one.

Moreover, the demonstration of a BD dose-response relationship in young children will suggest similarity between wheezy young children and older children and adults with asthma bronchial behaviour that may have possible therapeutic implications.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between 2 years 6 months and 6 years 11 months of age referred for pulmonary function testing with bronchodilator test, due to recurrent wheezing ,at least three times in the past year, to LFT laboratories at Armand Trousseau, Robert Debré, both in Paris and Arnaud de VILLENEUVE, in Montpellier hospitals
* No use of bronchodilator in the previous 12 hours before the test
* Parents gave their signed consent for the study

Exclusion Criteria:

Any patient aged 2 years 6 months and 6 years 11 months :

* with another chronic lung disease (bronchopulmonary dysplasia, chronic bronchitis, viral sequel, pathology of inhalation, thoracic-pulmonary malformation, tracheomalacia), anatomical or functional abnormality of the pharyngolaryngeal tract (tonsils touching or in contact with the uvula, laryngomalacia, subglottic stenosis, vocal cord paralysis, laryngeal obstruction)
* taking regular treatment including leukotrienes receptor antagonist during the week before the test.
* treated with oral glucocorticosteroids within 15 days before the test.
* without social security insurance
* with opposition of the family
* known intolerant to Salbutamol

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Estimate of bronchodilator dose-effect | 90 MINUTES
  Estimate of bronchodilator dose-effect in young children using the technique of interruption of airflow.

SECONDARY OUTCOMES:
Determine the minimum dose to be used routinely in a bronchodilator test and study the effect of environment on the dose-effect of the BD and the minimum dose to be used when testing the BD. | 90 minutes
  Determine the minimum dose of bronchodilator to use during a routine test to bronchodilator in young children to demonstrate bronchial reversibility.
  To study the effect of the environment (preventer treatment, atopy, disease control) on the BD dose-response relationship and the minimum BD dose to use to study bronchodilator response.
  Study on the genotype of the beta2-adrenergic receptor as a source of variation in the dose-response to bronchodilator.

CONTACTS AND LOCATIONS:
Overall Officials: Beydon Nicole, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Beydon, Paris, France

REFERENCES:
- [Result] Mukhopadhyay S, Seddon P, Earl G, Wileman E, Symes L, Olden C, Alberti C, Bremner S, Lansley A, Palmer CN, Beydon N. How can we optimise inhaled beta2 agonist dose as 'reliever' medicine for wheezy pre-school children? Study protocol for a randomised controlled trial. Trials. 2016 Nov 11;17(1):541. doi: 10.1186/s13063-016-1437-7. PMID 27836009
- [Result] Beydon N, Nguyen TT, Amsallem F, Denjean A, Fenu G, Seddon P, Mentre F, Alberti C, Lombardi E. Interrupter resistance to measure dose-response to salbutamol in wheezy preschool children. Pediatr Pulmonol. 2018 Sep;53(9):1252-1259. doi: 10.1002/ppul.24116. Epub 2018 Jul 3. PMID 29972634